CLINICAL TRIAL: NCT00339417
Title: Effect of Albendazole and Ivermectin Dose on Wuchereria Bancrofti Microfilarial Clearance in Mali: A Randomized, Open Label Study
Brief Title: Effect of Albendazole Dose on Clearance of Filarial Worms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Amy D. Klion, M.D./National Institute of Allergy and Infectious Diseases, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 999906107; 06-I-N107
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-08-17

CONDITIONS: Lymphatic Filariasis
Keywords: Lymphatic Filariasis; Chemotherapy
MeSH Terms: conditions — Elephantiasis, Filarial | interventions — Albendazole; Ivermectin

INTERVENTIONS:
Drug: Albendazole
Drug: Ivermectin

SUMMARY:
This study, conducted in Mali, West Africa, will determine whether a new treatment regimen for lymphatic filariasis can eliminate the disease more quickly than the standard regimen. Lymphatic filariasis is caused by infection with very small filarial worms called Wuchereria bancrofti that are spread by mosquitoes. The disease can cause swelling of the arms, legs, breast and genitalia and can progress to permanent swelling of the legs or arms called elephantiasis. Currently, patients in Mali are treated with a single dose of 400 mg of albendazole plus two doses of 200 mcg/kg of ivermectin each year. This study will use a regimen of 800 mg of albendazole twice a year plus 200 mcg/kg of ivermectin twice a year for 2 years. The study will see if the new regimen is more effective in lowering the numbers of Wuchereria bancrofti in the blood and will examine the effects of the two treatments on the adult worms living in the lymph system.

Healthy people between 14 and 65 years of age who live in the Mali village of N'Tessoni and are infected with Wuchereria bancrofti may be eligible for this study. Candidates are screened with a medical history, a brief physical examination and blood tests to check for infection with Wuchereria bancrofti and to measure white blood cell counts.

Participants undergo the following procedures:

-First visit

Ultrasound examination to look for filarial worms in the body.

Random assignment to receive either standard treatment or the experimental regimen

Urine pregnancy test for women of child-bearing age.

Receive first treatment dose.

-6-month visit

Short history, physical examination and blood test.

Second treatment dose for subjects in experimental treatment group.

Urine pregnancy test for women of childbearing age.

-1-year visit

Short history, physical examination and blood test.

Second or third treatment dose, depending on treatment group.

Repeat ultrasound in subjects whose first ultrasound detected adult worms.

Urine pregnancy test for women of childbearing age.

-18-month visit

Short history, physical examination and blood test.

Fourth treatment dose for subjects in experimental treatment group.

Urine pregnancy test for women of childbearing age.

-24-month visit

Short history, physical examination and blood test.

Repeat ultrasound in subjects whose first ultrasound detected adult worms.

Urine pregnancy test for women of childbearing age.

DETAILED DESCRIPTION:
Albendazole and ivermectin are currently used in combination for annual mass treatment of lymphatic filariasis in Africa. Although the drugs have been donated, the cost of such programs is very high and has proven to be a major impediment to the success of programs in many countries with limited financial resources. Data from albendazole treatment of other filarial infections and one study comparing single to multi-dose DEC/albendazole in lymphatic filariasis suggest that increased dose and/or frequency of albendazole dosing may be more effective in clearing microfilariae. Furthermore, the optimal dose of ivermectin for the treatment of lymphatic filariasis is greater than that being used in the current mass treatment program. In this study, 50 volunteers with microfilaremic Wuchereria bancrofti infection will be randomized to receive standard annual therapy (albendazole 400 mg + ivermectin 150 mcg/kg) or semiannual therapy with an increased albendazole dose (albendazole 800 mg + ivermectin 400 mcg/kg). If adequate numbers of microfilaremic subjects are recruited, an additional 25 volunteers will receive annual therapy with the increased dose combination. Microfilarial levels, as well as measures of adult worm burden (circulating antigen, ultrasound identification of adult worm nests) will be followed every six months for three years to assess the effects of the treatments.

ELIGIBILITY:
* INCLUSION CRITERIA (Screening):
* age 14 to 65.
* men and women*.

  * Please note: women are not permitted to leave their homes at night without the approval of their husband or, if they are not married, a parent or male guardian. Since this protocol involves blood drawing at night, such approval is necessary for participation.

EXCLUSION CRITERIA (Screening):

* non-volunteers.
* age less than 14 or greater than 65.
* pregnant by history.

INCLUSION CRITERIA (Treatment):

* age 14 to 65 years.
* men and women.*
* Wb microfilarial count greater than or equal to 50 mf/ml.

EXCLUSION CRITERIA (Treatment):

* non-volunteers.
* age less than 14 or greater than 65.
* pregnancy.
* Hgb less than 9 g/dl.
* Heavy alcohol use (more than 7 beer or other alcohol-containing drink/week).
* Temperature greater than 37.5C or other serious medical illnesses.
* history of benzimidazole allergy.
* history of ivermectin allergy.
* use of albendazole or ivermectin within the past 6 months.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2006-02-22; Primary Completion 2008-08-01 (Actual); Study Completion 2011-08-17 (Actual)

PRIMARY OUTCOMES:
Wb microfilarial levels | 12 months

SECONDARY OUTCOMES:
Adult worm burden as assessed by circulating antigen levels and visualization of worm nests by ultrasound | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bamako, Faculty of Medicine, Pharmacy and Odontostomatology, Bamako, Mali

REFERENCES:
- [Background] Beach MJ, Streit TG, Addiss DG, Prospere R, Roberts JM, Lammie PJ. Assessment of combined ivermectin and albendazole for treatment of intestinal helminth and Wuchereria bancrofti infections in Haitian schoolchildren. Am J Trop Med Hyg. 1999 Mar;60(3):479-86. doi: 10.4269/ajtmh.1999.60.479. PMID 10466981
- [Background] Addiss DG, Beach MJ, Streit TG, Lutwick S, LeConte FH, Lafontant JG, Hightower AW, Lammie PJ. Randomised placebo-controlled comparison of ivermectin and albendazole alone and in combination for Wuchereria bancrofti microfilaraemia in Haitian children. Lancet. 1997 Aug 16;350(9076):480-4. doi: 10.1016/S0140-6736(97)02231-9. PMID 9274584
- [Background] Horton J, Witt C, Ottesen EA, Lazdins JK, Addiss DG, Awadzi K, Beach MJ, Belizario VY, Dunyo SK, Espinel M, Gyapong JO, Hossain M, Ismail MM, Jayakody RL, Lammie PJ, Makunde W, Richard-Lenoble D, Selve B, Shenoy RK, Simonsen PE, Wamae CN, Weerasooriya MV. An analysis of the safety of the single dose, two drug regimens used in programmes to eliminate lymphatic filariasis. Parasitology. 2000;121 Suppl:S147-60. doi: 10.1017/s0031182000007423. PMID 11386686